CLINICAL TRIAL: NCT00852345
Title: Clofazamine in the Long Term Treatment of Leprosy, Phase III
Brief Title: Treatment Protocol for Clofazamine in the Long Term Treatment of Leprosy
Status: No longer available | Type: Expanded Access
Sponsor: Kaiser Permanente (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IRB 5347; KPSC IRB 5347 (Other: Kaiser Permanente)
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Leprosy
Keywords: multibacillary leprosy; leprosy; clofazamine
MeSH Terms: conditions — Leprosy; Leprosy, Multibacillary

INTERVENTIONS:
Drug: clofazamine — clofazamine 50mg po qday (duration varies according to physician)

SUMMARY:
Clofazimine has shown effectiveness in the treatment of leprosy for many years. The World Health Organization and the National Hansen's Disease Program consider clofazamine to be standard therapy for treatment of multibacillary leprosy. In recent years, the availability of the drug has become limited and is currently available only under a research protocol and is considered "investigational." Use of Clofazamine in patients presenting with lepromatous leprosy is necessary for patients exhibiting nerve involvement or lesions resistant to other therapies. This drug will be used prospectively for patients who require treatment of leprosy as deemed appropriate by a Kaiser Permanente Southern California physician.

DETAILED DESCRIPTION:
Treatment protocol objective is to treat patients with clofazamine who meet inclusion criteria stated above.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected leprosy confirmed by skin biopsy and/or slit skin smears.
* Multibacillary leprosy (lepromatous leprosy or borderline-lepromatous).
* Paucibacillary leprosy (borderline, borderline tuberculoid, or indeterminate) if there is involvement of the cranial nerves or active acute neuritis.
* Known or suspected ENL(erythema nodosum leprosum) (a specific immune reaction with painful skin nodules and fever)
* Known or suspected dapsone-resistant leprosy or relapsed leprosy.
* Intolerance of other antileprosy antibiotic (where clofazamine is substituted as apart of multidrug regimen)

Exclusion Criteria:

* Uncomplicated paucibacillary leprosy which would otherwise be treated with dapsone and rifampin only.
* Known prior intolerance of Clofazamine
* Any minor (even with parental consent)
* Any fertile woman who is pregnant a specific immune reaction with painful skin rash and fever)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Arnold M Henson, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente, Irvine, California, United States